CLINICAL TRIAL: NCT04227925
Title: The Longevity of Trichuris Trichiura Colonization
Status: Completed | Type: Observational
Sponsor: University of Aarhus (Other)
Responsible Party: Sponsor
Other Study IDs: T trichiura longevity
Record Dates: First submitted 2020-01-10; First posted 2020-01-14 (Actual); Last update posted 2020-01-14 (Actual); Status verified 2020-01

CONDITIONS: Helminthiasis; Helminth Infection
MeSH Terms: conditions — Helminthiasis; Trematode Infections | interventions — TT95 protein, Trichuris trichiura

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Biological: Trichuris trichiura — Infective eggs from human whipworm, Trichuris trichiura

SUMMARY:
The aim of the study was to study the longevity of Trichuris trichiura colonization

DETAILED DESCRIPTION:
The present study investigates the longevity of Trichuris trichiura colonization in a human volunteer as measured by regular fecal sampling.

ELIGIBILITY:
Inclusion Criteria:

The included volunteer is a researcher within parasitology with focus on Trichuris trichiura and Trichiura suis. He planned to infect himself under medical supervision. This was his third self-infection with Trichuris. The only clinical criterion for his inclusion in the study was that he was healthy.

Exclusion Criteria:

N/A

Ages: 18 Years to 70 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: A singlex healthy volunteer
Sampling Method: Non-Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2013-04-08 (Actual); Primary Completion 2019-09-17 (Actual); Study Completion 2019-09-17 (Actual)

PRIMARY OUTCOMES:
Faecal egg excretion | 78 weeks
  Regular monitoring of fecal egg counts by microscopy

IPD SHARING:
Plan to Share IPD: No